CLINICAL TRIAL: NCT06786611
Title: Enhanced Quantitative Assessment of Lumbar Facet Joint Degeneration: Refining the Weishaupt Grading System With Grayscale Curve Fitting and Imaging Parameter.
Brief Title: Quantitative Assessment of Lumbar Facet Joint Degeneration, A Retrospective Study.
Status: Completed | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024455; 2024DZXYY- 105 (Other: Shanghai Changzheng Hospital)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Facet Joint Pain; Low Back Pain; Facet Joints; Degeneration ; Deep Learning ;Artificial Intelligence; Facet Joint Disease
Keywords: facet joint degeneration; low back pain; Weishaupt grading system; Grayscale curve fitting
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- facet joint degeneration: based on the Weishaput grading system, we classified all included patients into the facet joint degeneration group and divided them into four subtypes according to different grades.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Based on the different manifestations of facet joints under MRI, and with the help of the characteristic manifestations of the gray value curve of facet joints under different subtypes, the curve of facet joints under the same level is fitted, and finally the accurate evaluation of different subtypes of small joints is achieved.

SUMMARY:
Observational study

The purpose of this observational study was to understand the quantitative assessment of the degree of degeneration of lumbar facet joints, and to improve the Weishaupt grading system by using gray-scale curve fitting and imaging parameters.

The main questions it aims to answer are: How to realize quantitative analysis of lumbar facet joint degeneration in patients with chronic low back pain with MRI?

The MRI information of patients with different grades of articular process joint degeneration has been statistically summarized in nearly 5 years

ELIGIBILITY:
Inclusion Criteria:

* (1) Age range from 20 to 80 years old; (2) Persisted chronic low back pain (CLBP) more than 12 weeks; (3) Complete preoperative X-ray and 1.5T MRI examination.

Exclusion Criteria:

* (1) Scoliosis, Cobb angle>20°; (2) Lack of preoperative X-ray or MRI examination; (3) 3.0T MRI; (4) The interval between preoperative X-ray and MRI examinations is more than one month; (5) Previous lumbar spine internal fixation surgery; (6) Lumbar spondylolisthesis > 5 mm, with severe dislocation of facet joints; (7) Intravertebral bone cement implantation; (8) Severe spinal joint disease (e.g. mandatory spondylitis); (9) Spinal tumors; (10) The maximum extension depth of Modic changes (MC) relative to vertebral body height was greater than 25%.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent imaging examination in Shanghai Changzheng Hospital from September 2020 to July 2024 to evaluate lumbar joint degeneration were included.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Grayscale Curve Fitting | "From enrollment to the end of treatment at 1 weeks
  Based on the signal intensity changes of T2-weighted of 1.5T MRI in different degenerative grades of facet joints, the gray value changes in facet joints were measured and fitted.

SECONDARY OUTCOMES:
Correlation analysis and logistic regression analysis between imaging parameters | "From enrollment to the end of treatment at 1 weeks
  Imaging parameters such as intervertebral space height (ISH), lumbar range of motion (ROM-L), intervertebral disc degeneration, facet joint degeneration, facet joint area, vertebral bone quality (VBQ) scores, subcutaneous fat tissue thickness (SFTT) and grayscale values of lumbar facet joint were analyzed. Statistical correlations were evaluated using spearman rank correlation and ordinal logistic regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
As the data involves the personal privacy of patients in our hospital, it is considered not to be published as public data. You can apply with the person in charge of this study for reasonable demands.